CLINICAL TRIAL: NCT06678685
Title: An Exploratory Study of Spironolactone Tablets for the Treatment of Children With NCOR Mutations
Brief Title: Spironolactone Improved Children With NCOR Mutations
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL000004
Record Dates: First submitted 2024-10-27; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: NCOR Gene Mutations; Spironolactone; ASD
MeSH Terms: interventions — Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- spironolactone treatment (Experimental)
  Interventions: Drug: .spironolactone

INTERVENTIONS:
Drug: .spironolactone — In the first week, the starting dose is 2mg/Kg per body weight once a day, taken with food at lunch every day, and subsequently adjusted according to the situation. If the patient's serum potassium is ≤5.0 mEq/L and the patient's serum creatinine is ≤2.5 mg/dL, treatment should be initiated with 25 mg spironolactone once daily. Increased to 100mg after remission. If the results are not obvious in the first month, increase the drug dose to 3mg/Kg.

SUMMARY:
NCOR1/2 constitutes the NCOR complex, which interacts with many different nuclear receptors to produce special physiological effects. These receptors further recruit epigenome modifying enzymes that are involved in the transcription of multiple genes involved in neurotransmission and synaptic plasticity. Studies of mice with gene knockout and autistic patients with NCOR mutations have found that both exhibit clinical symptoms characteristic of ASD, such as deficits in social interaction, spatial learning and impaired recognition memory. Further study revealed that the cause was the hyperexcitability of GABaergic neurons in the lateral hypothalamus (LH) due to the NCOR1/2 defect, which impaired synaptic plasticity in the hippocampal CA3 region through the single synaptic LHGABA-CA3 neural projection, and thus exhibited learning/memory impairment. Therefore, drugs that affect the NCOR receptor can improve learning/memory impairment by affecting GABA neurons. Spironolactone is a widely used diuretic with good safety. It is widely used in the treatment of hypertension, edema and anti-androgen therapy in children. In this study, spironolactone is one of the most popular drugs used to treat children with NCOR gene mutation. In our previous animal experiments, we found that spironolactone could treat NCOR mutant mice and improve ASD-related symptoms, such as reduced sensorimotor capacity, learning disability and impaired working memory; Moreover, the efficacy of related diuretics in the treatment of ASD diseases has been proved clinically. So spironolactone may be a new target for the treatment of NCOR patients in the future.

ELIGIBILITY:
Inclusion Criteria:

1. ADOS-2 diagnostic criteria for autistic children
2. Patients with NCOR1/2 gene mutation detected by whole exon test;
3. Age: 3-10 years old;
4. The subject and (or) guardian sign the informed consent, agreeing that the researcher will cooperate with the clinical trial process and collect clinical data and peripheral blood and urine samples;

Exclusion Criteria:

1. have other pathogenic mutations (confidence higher than the NCOR1/2 mutation);
2. Boys over 10 years old;
3. Allergic to spironolactone, used spironolactone one month before enrollment;
4. Hyperkalemia, serum potassium concentration > 5.5mmol/L;
5. Renal insufficiency;
6. Used related drugs one month before enrollment: potassium supplement, angiotensin-converting enzyme inhibitor, angiotensin receptor blocker, digoxin, coletenamine, acetylsalicylic acid, abiraterone;
7. Fever (body temperature above 37.3°);
8. Clinically significant metabolic, hematological, liver, immune, urological, endocrine, neurological, pulmonary, psychiatric, skin, allergic, renal, or other major conditions in the determination of ASD that may affect the interpretation of study findings or patient safety.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Wechsler Intelligence Scale for Children, Fourth Edition (WISC-IV) | 1. Baseline 2. At the end of Cycle 1 (each cycle is 60 days) 3.At the end of Cycle 2 (each cycle is 60 days)
  Scores range from 40 to 130, with higher scores representing higher intelligence
Autism Diagnostic Observation Scale-2 | 1. Baseline 2. At the end of Cycle 1 (each cycle is 60 days) 3.At the end of Cycle 2 (each cycle is 60 days)
  The score ranges from 0 to 9, with higher scores indicating more severe autism
The amount of gamma amino butyric acid(GABA) in brain | 1. Baseline 2. At the end of Cycle 1 (each cycle is 60 days) 3.At the end of Cycle 2 (each cycle is 60 days)

SECONDARY OUTCOMES:
Blood pressure | 1. Baseline 2. At the end of Cycle 1 (each cycle is 60 days) 3.At the end of Cycle 2 (each cycle is 60 days)
  Including systolic and diastolic blood pressure
The Score of Developmental Neuropsychological Assessment(NEPSY-2 Scale ) | 1. Baseline 2. At the end of Cycle 1 (each cycle is 60 days) 3.At the end of Cycle 2 (each cycle is 60 days)
  Scores range from 0 to 100, with higher scores representing stronger neurodevelopment